CLINICAL TRIAL: NCT07138794
Title: Ultrasound-Guided Subtransverse Interligamentary Block Versus Thoracic Paravertebral Block for Postoperative Analgesia in Patients Undergoing Open Nephrectomy: A Randomized Clinical Trial
Brief Title: Ultrasound-Guided Subtransverse Interligamentary Block Versus Thoracic Paravertebral Block for Postoperative Analgesia in Patients Undergoing Open Nephrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR1283/7/25
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Subtransverse Interligamentary Block; Thoracic Paravertebral Block; Postoperative Analgesia; Open Nephrectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STIL group (Experimental): Patients will receive subtransverse process interligamentary (STIL) block using 20ml of bupivacaine 0.25%.
  Interventions: Other: Subtransverse process interligamentary
- TPVB group (Experimental): Patients will receive a thoracic paravertebral block (TPVB) using 20ml of bupivacaine 0.25%.
  Interventions: Other: Thoracic paravertebral block

INTERVENTIONS:
Other: Subtransverse process interligamentary — Patients will receive subtransverse process interligamentary (STIL) block using 20ml of bupivacaine 0.25%.
  Arms: STIL group
Other: Thoracic paravertebral block — Patients will receive a thoracic paravertebral block (TPVB) using 20ml of bupivacaine 0.25%.
  Arms: TPVB group

SUMMARY:
This study aims to compare ultrasound-guided subtransverse process interligamentary (STIL) block versus thoracic paravertebral block (TPVB) for postoperative analgesia in patients undergoing open nephrectomy.

DETAILED DESCRIPTION:
Acute pain physiopathology is explained as it is mediated by inflammatory cell infiltration, activation of spinal cord pain pathways, and also by reflexive muscle spasm. All of these three mechanisms of acute pain are typically ameliorated during the postoperative recovery.

A thoracic paravertebral block (TPVB) shows comparable analgesic efficacy with fewer side effects compared with thoracic epidural analgesia in patients undergoing thoracotomy.

The recently introduced subtransverse process interligamentary (STIL) block offers a safer alternative by targeting thoracic nerves without entering paravertebral space.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-III.
* Undergoing open nephrectomy under general anesthesia.

Exclusion Criteria:

* History of allergies to local anesthetics.
* Opioid dependency.
* Bleeding or coagulation disorders.
* Psychiatric and neurological disorder.
* Local infection at the site of injection.
* Body mass index (BMI) > 35 kg/m2.
* Severe heart, lung, liver, and renal dysfunction.
* Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-08-23 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption | 48 hours postoperatively
  Rescue analgesia of morphine will be given as 3 mg bolus if the numeric rating scale (NRS) > 3 to be repeated after 30 min if pain persists until the NRS < 4.

SECONDARY OUTCOMES:
Time to the 1st rescue analgesia | 48 hours postoperatively
  Time to the first request for the rescue analgesia will be recorded from the end of surgery to first dose of morphine administrated.
Intraoperative fentanyl consumption | Intraoperatively
  Additional fentanyl bolus dosages of 0.5 µg/kg IV will be administered if heart rate or mean arterial blood pressure elevated more than 20% of the baseline (after exclusion of other causes than pain).
Mean arterial pressure | Till the end of surgery (Up to 2 hours)
  Mean arterial pressure will be recorded preoperatively, before performing the block, and every 15 min till the end of surgery.
Heart rate | Till the end of surgery (Up to 2 hours)
  Heart rate will be recorded preoperatively, before performing the block, and every 15 min till the end of surgery.
Degree of pain | 48 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the numeric rating scale (NRS) score. NRS (0 represents "no pain" while 10 represents "the worst pain imaginable"). NRS will be assessed at PACU, 2, 4, 6, 8, 12, 18, 24, 36, and 48 h postoperatively.
Incidence of adverse events | 48 hours postoperatively
  Incidence of adverse events such as pneumothorax, local anesthetic systemic toxicity (LAST), bradycardia, hypotension, nausea, vomiting, respiratory depression, pruritus, or any other complication will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.